CLINICAL TRIAL: NCT05451745
Title: Incidence of and Risk Factors for Glaucoma Following Pediatric Cataract Surgery: 10 Years Longitudinal Study
Brief Title: Glaucoma Following Pediatric Cataract Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: CCMPOH2022
Record Dates: First submitted 2022-06-26; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma Following Pediatric Cataract Surgery; Glaucoma Secondary; Congenital Cataract
Keywords: Pediatric Cataract; Congenital Cataract; Glaucoma following cataract surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to report the incidence and related risk factors glaucoma following cataract surgery (GFCS). and to provide evidence-based evidence for the development of standardized follow-up methods or diagnosis and treatment decisions.

DETAILED DESCRIPTION:
A secondary clinical data analysis from a prospective longitudinal cohort study. A total of 819 children with congenital cataracts (CC) were included from January 2011 to December 2016, and the follow-up deadline was January 31, 2022. All study subjects were under 18 years old, and the average follow-up time after cataract extraction was over 5 years. The children were divided into subgroups according to whether the intraocular lens (IOL) was implanted or not after cataract surgery, and the clinical characteristics were compared. Cox regression analysis model and Kaplan-Meier survival analysis model were used to investigate the incidence, cumulative risk probability and related risk factors of GFCS events. A nomogram was used to build a predictive model for the occurrence of GFCS.

ELIGIBILITY:
Inclusion Criteria:

* 1) The guardian of the child voluntarily signed the informed consent;
* 2) The age is ≤18 years old, and the gender is not limited;
* 3) The diagnostic criteria for congenital cataract are met; the lens is opacified in one or both eyes;
* 4) The intraocular pressure before cataract extraction is normal ( less than 21 mmHg, considering the errors caused by different intraocular pressure measurement methods and different anesthesia methods);
* 5) The children have no glaucoma-related clinical manifestations and signs before cataract extraction, such as large corneal diameter, corneal edema or opacity, Increased cup-to-disk ratio, etc.;
* 6) The child has no family history of glaucoma;
* 7) Cataract extraction was performed in our hospital, and/or no intraocular lens was implanted;
* 9) Clinical diagnosis of glaucoma following cataract surgery
* 10) The postoperative follow-up time was not less than 60 months.

Exclusion Criteria:

* 1) Have received other eye surgery before enrollment, including cataract surgery, anti-glaucoma surgery, and corneal surgery, etc.;
* 2) Combined with congenital glaucoma, a clear history of eye trauma, and other complex eyes medical history (including persistent Persistent hyperplastic primary vitreous (PHPV), Peter's anomaly, congenital aniridia, Marfan syndrome, lens insufficiency, retinitis pigmentosa, high myopia, fundus lesions, congenital rubella syndrome, ocular brain-renal syndrome
* 3) Combined with other serious systemic diseases (cardiovascular, respiratory, digestive, urinary, nervous, and other system diseases)

Clinical diagnosis of glaucoma following cataract surgery:

after cataract removal, two or more of the following are required

1. Intraocular pressure: >21 mmHg (investigator discretion on the method of measurement and if EUA (Examination Under Anesthesia) data alone is sufficient).
2. Visual fields: reproducible visual field defect that is consistent with glaucomatous optic neuropathy with no other observable reason for the visual field defect.
3. Axial length: progressive myopia or myopic shift with increased ocular dimensions that outpace normal growth.
4. Cornea: findings including Haab striae, corneal diameter >11mm in newborns, >12mm in children younger than 1 year old, and >13mm in children older than 1 year old.
5. Optic nerve: progressive increase in the cup-disc ratio, cup-disc asymmetry of 0.2 when optic discs are of similar size, and focal rim thinning.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Relying on the congenital cataract research platform established by our hospital, this prospective cohort clinical study will prospectively register children with congenital cataracts who underwent cataract extraction in our hospital from January 2010 to December 2016.
Sampling Method: Probability Sample
Enrollment: 819 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of glaucoma following congenital cataracts | up to 10 years
  A Kaplan-Meier analysis was used.
Risk factors of glaucoma following cataract surgery | up to 10 years
  To use Cox regression analysis to evaluate the potential risk factors in GFCS.

REFERENCES:
- [Background] Lin H, Chen W, Luo L, Zhang X, Chen J, Lin Z, Qu B, Zhan J, Zheng D, Zhong X, Tian Z, Liu Y; Study Group of CCPMOH. Ocular hypertension after pediatric cataract surgery: baseline characteristics and first-year report. PLoS One. 2013 Jul 29;8(7):e69867. doi: 10.1371/journal.pone.0069867. Print 2013. PMID 23922832
- [Background] Wang J, Chen J, Chen W, Wang Q, Zhao L, Wang R, Liu Z, Chen H, Cao Q, Tan X, Lin Z, Li X, Li J, Lai W, Zhu Y, Chen C, Zheng D, Wu M, Han Y, Chen W, Liu Y, Lin H. Incidence of and Risk Factors for Suspected Glaucoma and Glaucoma After Congenital and Infantile Cataract Surgery: A Longitudinal Study in China. J Glaucoma. 2020 Jan;29(1):46-52. doi: 10.1097/IJG.0000000000001398. PMID 31688374